CLINICAL TRIAL: NCT01855360
Title: An 18 Month, Open Label Study of the Tolerability and Efficacy of a Combination of Doxycycline and Tauroursodeoxycholic Acid (TUDCA) in Patients With Transthyretin Amyloid Cardiomyopathy.
Brief Title: Doxycycline and TUDCA in Patients With Transthyretin Amyloid Cardiomyopathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Rodney H. Falk, MD, Director, Brigham and Women's Hospital Cardiac Amyloidosis Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BWHAMY1
Record Dates: First submitted 2013-03-12; First posted 2013-05-16 (Estimated); Results first posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2018-11

CONDITIONS: Amyloidosis; Heart (Manifestation); Senile Cardiac Amyloidosis
Keywords: amyloid; amyloidosis; cardiac amyloidosis; senile amyloidosis; familial amyloidosis; transthyretin amyloidosis
MeSH Terms: conditions — Amyloidosis; Amyloid Neuropathies, Familial; Alzheimer Disease; Amyloidosis, Familial; Amyloidosis, Hereditary, Transthyretin-Related | interventions — ursodoxicoltaurine; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TUDCA and Doxycycline (Experimental): INTERVENTION: Patients meeting study criteria were prescribed TUDCA taken orally, 250 mg three times daily. and doxycycline taken orally, 100 mg twice daily.
  Interventions: Drug: Tauroursodeoxycholic Acid and Doxycycline

INTERVENTIONS:
Drug: Tauroursodeoxycholic Acid and Doxycycline
  Other Names: Doxycycline:Vibramycin, Monodox, Acticlate, Atridox, Avidoxy, Doxy, Doxycin, Doryx, Oracea, Periostat, Adoxa, Ocudox, and Doryx MPC.

SUMMARY:
The objective of the study is to determine whether the combination of the bile acid TUDCA, and doxycycline will slow the progression of familial and senile amyloidosis.

DETAILED DESCRIPTION:
Primary objectives The study is designed to prospectively evaluate the efficacy of doxycycline and TUDCA, prescribed together, on cardiac disease progression in patients with senile systemic amyloidosis or familial amyloidosis due to a TTR mutation. The definition of progression will be defined, primarily, by echocardiographic indices , as well as by serial cardiac biomarkers, specifically NT-proBNP.

. Echocardiographic details

. Standard parameters of wall thickness, chamber size, Doppler echocardiographic assessment of valvular function and diastolic function will be measured.

The primary endpoint is the response rate to doxycycline + TUDCA treatment at month 12 and 18, based upon echocardiographic findings. Since the precise echocardiographic findings will determine the definition of a responder, an approximate figure on which progression is based will be given here, based on our previous, preliminary data. A responder will be defined as a patient with echocardiographic evidence of stability of speckle strain parameters at 12 months of therapy with doxycycline/TUDCA. Based on our preliminary work, this is currently defined as a change in absolute longitudinal strain of < -2%, but the use of this parameter may alter slightly after the part 1 analysis.

Secondary endpoints

Secondary endpoints of the study are:

* to assess the tolerability and safety of the treatment, based on evaluation of the development of recognized side-effects, such as photosensitivity, drug sensitivity, gastrointestinal disturbance and superinfection, as well as any other unexpected effects potentially attributed to therapy.
* to assess change from baseline in QoL (SF-36 scale) at months 6, 12 and 18;

This is an 18-month, open label treatment period in which doxycycline (100 mg twice daily) and TUDCA (250 mg, three times daily) are administered to 30 consenting subjects with SSA amyloidosis and 10 subjects with ATTR amyloidosis. Subjects will be evaluated at baseline, and then after 6, 12, and 18 months of doxycycline plus TUDCA treatment or at time of premature treatment discontinuation. Monthly phone contacts and regular blood tests will be performed to monitor potential adverse events.

All eligible subjects will receive doxycycline hyclate (100 mg twice daily) as well as TUDCA 250 mg three times a day orally. Treatment will be initiated with doxycycline 100 mg daily for 1 week, to assess tolerance, and then increased to twice daily for week 2, following which repeat blood tests of BUN, creatinine , electrolytes and liver function tests will be drawn. If these are stable, TUDCA will be added at the above dose, and the combination will be administered for 17.5 months. TUDCA, formulated in capsules of 250 mg, will be provided at enrolment and at subsequent study visits. Doxycycline will be prescribed through the patient's own pharmacy as it is a widely available drug and is already being used as a single agent in some patients with cardiac amyloidosis (including in our own program).

In patients in whom doxycycline is poorly tolerated due to gastrointestinal symptoms and/or mild, transient reduction in blood cell counts, the treatment schedule will be modified according to the protocol of Obici et al and doxycycline will be administered cyclically (200 mg/day for 28 days every six weeks up to 18 months). In these patients TUDCA will continue to be administered at 250 mg, three times daily.

The following study procedures will be performed at scheduled visits. Entry evaluation

After obtaining consent, subjects will undergo:

1. Physical examination
2. ECG
3. Quality of Life questionnaire (SF-36)
4. A full echocardiographic study (standard clinical practice)
5. Serum creatinine, AST, ALT, total bilirubin, CBC, NT-proBNP, troponin I, alkaline phosphatase, and pregnancy test (if applicable)

6-monthly visits

Every 6 months subjects will follow-up with the Investigator for standard blood work and physical examination, to evaluate tolerability of the treatment, and to have an echocardiogram. ) .

Phone contacts 3-Monthly phone contacts between clinic visits will be performed by the research coordinator for monitoring of the treatment safety. to the IRB, as per IRB regulations.

Echocardiograms will be read blindly to determine standard echocardiographic parameters, with an emphasis on those that may change in progressive cardiac amyloidosis (LV mean wall thickness, quantitative LV ejection fraction, LV dimensions etc)..

Study Endpoints Response will be evaluated at Month 12 by means of the percentage of subjects with stability in echocardiographic parameters, as initially defined based on the 40 patients studied by serial echocardiography. Analysis will be performed both as an evaluation of the percentage of the group whose cardiac function remains stable, and as an analysis of the mean change in echocardiographic parameters compared to the historical control group. Details of the drug regimen tolerability will also be analyzed. Patients will continue in the study for an additional 6 months (duration of treatment 18 months) with a repeat (secondary) analysis of the same parameters at 18 months (secondary endpoint).

.

Subjects discontinuing study participation prematurely due to drug intolerance will, if agreeable, undergo a full Study Site visit evaluation. This assessment will include the routine 6-montly tests, with the exclusion of a repeat echocardiogram if one has been done in the past 4 months.

Efficacy observations and measurements For efficacy evaluation, subjects will be interviewed and examined every 6 months. Echocardiograms, obtained at 0, 6, 12 and 18 months will be analyzed for standard measurements as well as by strain imaging using a dedicated Echo-Pac analysis system. Cardiac biomarkers will be obtained every 6months.

SF-36 Quality of Life questionnaires will be administered at baseline and 6, 12, and 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented transthyretin cardiac amyloidosis by biopsy and staining using immunohistochemistry or mass spectrometry
* Echocardiographic appearance of left ventricular wall thickness of 13mm or more in the absence of hypertensive heart disease
* Confirmed ATTR or SSA by genetic testing
* Age 18-90
* Male or non-pregnant, non-lactating females
* Willingness to return to the treatment center for follow-up

Exclusion Criteria:

* Prior liver transplantation or liver transplantation anticipated in less than 6 months
* Alanine Transaminase and/or Aspartate Transaminase ≥2 x upper normal limit (UNL)
* Alkaline Phosphatase ≥2 x UNL
* Creatinine clearance <20 mL/min
* Any other lab values that in the opinion of the investigator might place the subject at unacceptable risk for participation in the study
* History of poor compliance
* History of hypersensitivity to any of the ingredients of the study therapies
* Any investigational drug within 4 weeks prior to study entry or during the study
* Current use of diflunisal for therapy of amyloidosis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2015-05-31 (Actual); Study Completion 2015-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rodney H Falk, MD, Principal Investigator — Brigham and Women's Hospital, Boston MA
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- TUDCA and Doxycycline: INTERVENTION: Patients meeting study criteria were prescribed TUDCA taken orally, 250 mg three times daily. and doxycycline taken orally, 100 mg twice daily.
  Tauroursodeoxycholic Acid and Doxycycline
Period: Overall Study
Arm/Group | TUDCA and Doxycycline
Started | 40
Completed | 30
Not Completed | 10

BASELINE CHARACTERISTICS:
Arm/Group | TUDCA and Doxycycline
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Number analyzed is number of patients completing 12 month visit and who had a technically analyzable echocardiogram.
  years
    number analyzed (Participants) | 30
    (all) | 71.3 (3.5)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Number analyzed is number of patients completing 12 month visit and who had a technically analyzable echocardiogram (this was the primary endpoint).
  Participants
    number analyzed (Participants) | 30
    Female | 1
    Male | 29
Region of Enrollment [Count of Participants; unit: Participants] — Population: Number analyzed is number of patients completing 12 month visit and who had a technically analyzable echocardiogram.
  Participants
    United States: number analyzed (Participants) | 30
    United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Changes in Strain Echocardiography
Description: Outcome measure, namely changes in longitudinal echocardiographic strain, will be compared to previously determined changes derived from a cohort of patients with TTR cardiac amyloidosis who were not receiving specific therapy for amyloid deposition.
Time Frame: Time Frame: * (FDAAA) outcome measure is assessed every 6 months by serial echocardiography, with final measurement 18 months after enrollment, change at 12 months reported as pre-defined primary endpoint.
Population: Patients who completed 18 month visit (primary outcome) and had a technically adequate echocardiogram to analyze strain imaging
Measure: Mean (Standard Deviation); unit: percent LV shortening
Arm/Group | TUDCA and Doxycycline
Number analyzed (Participants) | 30
percent LV shortening | 9.1 (.9)

2. Secondary Outcome: Number of Patients With Adverse Events
Time Frame: 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | TUDCA and Doxycycline
Number analyzed (Participants) | 40
Participants | 7

ADVERSE EVENTS:
Time Frame: Adverse events collected over the course of 18 months.
Arm/Group | TUDCA and Doxycycline
All-Cause Mortality (participants affected / at risk) | 6/40
Serious Adverse Events (participants affected / at risk) | 1/40
Other Adverse Events (participants affected / at risk) | 6/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TUDCA and Doxycycline (N=40)
acute kidney injury (Renal and urinary disorders) | 1 (1) — 1 patient developed worse renal function on drug, with heart block. Unclear whether worsening renal function was due to low cardiac output caused by heart block (i.e progression of disease) or whether drug combination aggravated renal function.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TUDCA and Doxycycline (N=40)
gastrointestinal upset (Gastrointestinal disorders) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes